Version Number: V1.0

Date: August 31, 2018

## Study Protocol

A Multicenter prospective cohort study on the risk factors for gallbladder cancer

Researcher: Wang Jianming

Research institute: Huazhong University of Science

Tongji Hospital, Tongji Medical College

Date: August 31, 2018

# Study Protocol Summary

| Title | A Multicenter prospective cohort study on the risk factors for gallbladder cancer |
|---|---|
| Research Institute | Huazhong University of Science Tongji<br>Hospital, Tongji Medical College |
| Number of research Institute | 220 |
| Research Purposes | 1. To study the correlation between benign gallbladder disease and gallbladder cancer; |
| | 2. Explain the timing of intervention for benign gallbladder disease, the mode of intervention, and the benefits of early prevention of gallbladder cancer, and further calculate the difference in socioeconomic benefits (the cost of medical care caused by the disease). |
| Research Design | Prospective, multi-centred research |
| Sample size determination basis | This trial is a prospective study, the main purpose of the study is to investigate the association between benign gallbladder disease and gallbladder carcinoma; to explain the timing of intervention, intervention and early prevention of benign gallbladder disease; according to the national epidemiology of gallbladder cancer Center Clinical Research (unpublished), 2000 National Cholecystoma Clinical Epidemiology Report, and 2005 Clinical Analysis of 2379 Cases of Gallbladder Carcinoma in 17 Hospitals in Five Northwest Provinces, Preexperimental data, using samples The volume estimation formula, $\alpha = 0.05$ , $\beta = 0.1$ , plans to enroll 100,000 people. |

| Standard constrain | Subjects who met the following four criteria entered the study. (1) A benign gallbladder disease (according to any imaging test result) during a physical examination or visit; (2) healthy people without gallbladder disease; (3) Age greater than 18 years and less than 80 years old; (4) Sign the informed consent form. |
|---|---|
| Exclusion criteria | Subjects can not enter the study by combining any of the following (1) Concomitant diseases such as severe mental illness, severe heart, lung and kidney; (2) Refusal of follow-up requirements. |
| Observation index | <ul> <li>(1) Incidence of gallbladder cancer;</li> <li>(2) Gallbladder-related disease mortality;</li> <li>(3) Gallbladder-related disease surgery rate;</li> <li>(4) Gallbladder related diseases surgery;</li> <li>(5) Medical expenses for gallbladder related diseases;</li> </ul> |
| Research period | 3 years |
| Statistical analysis | The Linklab information collection system is used for data entry and verification. All data was counted using SPSS 21.0. |

# Table

| Background | 1 |
|----------------------------------------------|----|
| 二、 Purpose | 2 |
| 三、 Content | 2 |
| 3.1 Research Type | 2 |
| 3.2 Population | 2 |
| 3.2.1 Inclusion criteria | 2 |
| 3.2.2 Exclusion criteria | 2 |
| 3.2.3 Exit case | 2 |
| 3.2.4 Treatment of withdrawal cases | 3 |
| 3. 2. 5Group | 3 |
| 3.3 Grouping Method | 3 |
| 3. 4Procedures | 3 |
| 3.4.1Research Period | 3 |
| 3. 4. 2Recruitment | 3 |
| 3. 4. 3 Follow-up | 4 |
| 3.4.4 Observation Index | 4 |
| 四、Statistical analysis | 4 |
| 4.1 Sample size estimation | 4 |
| 4.2 Statistics and Analysis of Research Data | 5 |
| 五、 Research on related ethics | 5 |
| 5.1 Audit by Ethics Committee | 5 |
| 5. 2Consent Form | 6 |
| 六、 Confidentiality Measures | 6 |
| 七、 Researcher | |
| 7.1 Research Institute | 7 |
| 7.2Participants | 12 |
| 八、Reference | 13 |

## 一、Backgroud

Gallbladder cancer is the most common malignant biliary tract neoplasm. The incidence of gallbladder cancer is increasing year by year, ranking sixth in the incidence of digestive tract cancer. [1] There are significant differences in the incidence of gallbladder cancer globally. It has been reported that the incidence of gallbladder cancer varies 25 times in different regions. The reasons for this difference may be related to environmental exposure differences and inherent genetic susceptibility. The highest incidence was found in the Andes Mountains of South America, Eastern and Central Europe (such as Hungary, Germany and Poland), Israel, while the incidence was lower in the United States and most Western and Mediterranean countries (such as Britain, France and Norway). In Asia, the incidence of gallbladder cancer is also at a high level, especially among women and men in northern India and Pakistan, while Korea has the highest incidence in Asia. The incidence of primary gallbladder cancer in China accounted for 0.4%-3.8% of biliary tract diseases in the same period, and there were regional differences. [2].

The main risk factors of gallbladder cancer include gallstone, gallbladder polyp, gallbladder adenoma, chronic inflammation of gallbladder, etc. [3][4]. However, in recent years, there is still lack of relevant risk factors evaluation data, so on the basis of large-scale epidemiological investigation, large-scale prospective research is needed to further clarify the level of risk factors related to gallbladder cancer.

With the development of modern imaging technology and indepth understanding of gallbladder diseases, the detection rate of benign lesions of gallbladder (gallbladder polyps, gallbladder adenomyosis, gallbladder adenoma, gallbladder stones, etc.) is increasing year by year, while some benign lesions of gallbladder can gradually evolve into gallbladder cancer through a series of pathophysiological processes. Radical resection is the only possible method to cure or improve the long-term survival rate of gallbladder cancer. However, due to the difficulty in early diagnosis of gallbladder cancer, the unknown etiology and lack of specific clinical manifestations, most patients were found to be advanced, with low resection rate and insensitive to radiotherapy and chemotherapy. [7] Most patients have lost the chance of operation at the time of consultation, and the overall 5-year survival rate is less than 5%. [5][6]. In the early stage of gallbladder cancer, because the biliary surgeon is not clear about the standard of standardized operation, the recurrence and metastasis of gallbladder cancer occur soon after operation, which seriously affects the prognosis [8]. Therefore, the correct understanding of benign gallbladder diseases, intervention time and intervention measures have always been a serious challenge for surgeons.

Correct understanding of the relationship between benign lesions of gallbladder and gallbladder cancer and rational grasp of the timing of surgical treatment are the urgent needs of many clinicians.

The purpose of this study was to establish a prospective cohort of benign gallbladder diseases and to explore the correlation between benign gallbladder diseases and gallbladder cancer, the timing of intervention and socioeconomic benefits. In order to further understand the epidemiological trend, diagnosis and treatment of benign gallbladder diseases in China, the Biliary Surgery Group of the Surgical Society of the Chinese Medical Association plans

to launch a nationwide epidemiological survey of gallbladder cancer (2018). This study will provide a more detailed basis for the diagnosis and treatment of benign gallbladder diseases in China.

## 二、Purpose

- 1. To study the correlation between benign diseases of gallbladder (such as gallstone, gallbladder polyp, gallbladder adenoma, cholecystitis, etc.) and gallbladder cancer:
- 2. To clarify the intervention timing, intervention methods and benefits of early prevention of gallbladder cancer for benign gallbladder diseases, and to further calculate the difference of socioeconomic benefits (medical costs caused by diseases).

#### 三、Content

#### 3. 1 Type

Prospective, multi-centred research

#### 3.2 Population

- (1) Patients with benign gallbladder diseases
- (2) Healthy people without gallbladder disease

#### 3.2.1 Inclusion Criteria

The subjects entered the study if they met the following four criteria.

- (1) Benign diseases of gallbladder were found during physical examination or consultation (according to the results of any imaging examination);
  - (2) Healthy people without gallbladder disease;
- (3) older than 18 years old and younger than 80 years old;

(4) Sign the informed consent.

#### 3.2.2 Exclusion criteria

If any of the following items are combined, participants will not be able to enter the study.

- (1) Complicated with severe mental illness, severe heart, lung and kidney diseases;
  - (2) Refusal of follow-up requests.

#### 3.2.3 Exit case

#### (1) Judgment

No matter when and why they quit, as long as they have not completed the whole follow-up observation, they are considered as cases of Midway withdrawal.

#### (2) Standard

- 1) Withdrawal from the study due to adverse events;
- 2) Serious breach of the plan;
- 3) Patients withdraw their informed consent.
- 4) Researchers believe that subjects need to quit.
- 5) others;

## 3.2.4 Management

Detailed records of withdrawal cases have been followed up, and statistical analysis of its observation indicators, the source documents should be kept for reference. Withdrawal rate should not exceed 20% during follow-up.

## 3.2.5 Group

Non exposed group: Healthy people without gallbladder disease

Exposed group: Imaging examination confirmed gallbladder disease (non-gallbladder cancer).

### 3.3 Number of cases and grouping method

This study is an observational study. There is two groups of subjects and 100,000 cases are planned to be enrolled.

#### 3.4 Research procedures and related examinations

#### 3.4.1 Research period

Case entry period:

All clinical research centers completed case collection within 20 years after the start of the study.

#### 3.4.2 Formulate CRF table and recruitment

- 1) Collect the information of patients: general demographic data; current medical history, past medical history, occupational history, residence history, personal habits, diet history, etc; imaging examination, blood routine, biochemistry, liver and kidney function, coagulation function, tumor markers and urine routine tests, routine preoperative examination (abdominal color Doppler ultrasound, CT, MR). Medical expenses related to diseases (including medical treatment, treatment, transportation, missed work, etc.).
- 2) Recruited subjects can be enrolled into the group after they have informed the patient about the research and signed the informed consent form of the clinical study; the relevant information of patients is recorded in the data collection form.

#### 3. 4. 3 Follow-up

#### (1) Follow-up period

Subjects were followed up once a year after they entered the queue. Outpatient, home or telephone follow-up was conducted. Understand the general situation of the subjects, laboratory examination results, radiological examination results, treatment and so on.

#### (2) Follow-up Protocol

- 1) Follow-up staff: Attending and special follow-up staff
- 2) Follow up mode: Outpatient, door-to-door or telephone follow-up.
- 3) Follow-up period: 20 years
- 4) Follow-up content: Collect information according to the main content of CRF table.
- 5) Follow-up End: ①Gallbladder tumor;
  - 2Dead;
  - 3 Acceptance of cholecystectomy.

#### 3.4.4 Observation index

- (1) Incidence of gallbladder cancer:
- (2) Mortality of gallbladder-related diseases;
- (3) Surgical rate of gallbladder-related diseases;
- (4) Surgical methods for gallbladder-related diseases;
- (5) Medical expenses for gallbladder-related diseases.

## 四、Statistical Analysis

## 4.1 Sample size estimation

- (1) Patients who meet the discharge criteria should be admitted to the group continuously without selectivity.
- (2) This experiment is an observational study. The main purpose of this study is to study the correlation between benign diseases of gallbladder (such as gallstone, gallbladder polyp, gallbladder adenoma, cholecystitis, etc.)

and the occurrence of gallbladder cancer, to clarify the timing, mode of intervention for benign diseases of gallbladder and the benefits of early prevention of gallbladder cancer, and to further calculate its socioeconomic Benefit difference (medical cost caused by disease). The incidence of gallbladder cancer was calculated according to the data of the previous "National Multicenter Clinical Study of Gallbladder Cancer Epidemiology" (unpublished), 2000 "National Clinical Epidemiological Investigation Report of Gallbladder Cancer" and 2015 "Clinical Analysis of 2379 Cases of Gallbladder Cancer in 17 Hospitals of Northwest Five Provinces". Calculate, use the sample size estimation formula,  $\alpha = 0.05$ ,  $\beta = 0.1$ , estimate the sample size of 100,000 people.

## 4.2 Data statistics and analysis

#### (1) Statistical grouping

- The patients were grouped according to their basic information and tabulated, such as:
  - Age: 01d (>60 years) , Middle-aged (45-59 years) , Youth (<=45)
    - Sex: Male, Female
- Location: According to the province where the patient is located
- History of present illness: Time of consultation, time of onset, symptoms of consultation, signs of admission, etc.
- Anamnesis: According to the past medical history, it can be divided into: biliary tract diseases (gallstones, gallbladder polyps), tumors, cardiovascular diseases, surgical history, etc.

• • • • • • • •

- (2) Statistics and Analysis of Research Data
  Linklab information acquisition system is used to input
  and verify data. All data were collected by SPSS 21.0. The
  data were analyzed by conventional single factor statistical
  analysis and advanced statistical methods (using CMH chisquare on demand, multifactor generalized linear regression,
  tendency score, etc.).
- (3) For the missing values of the main evaluation indicators, Multi-Filling method is used to correct and sensitivity analysis.
  - (5) Summary statistics
- Metrological data give mean, standard deviation, minimum, maximum, P25, median and P75; Counting data give frequency distribution and corresponding percentage.

#### 五、Research on Related Ethics

#### 5.1 Audit by Ethics Committee

This clinical study must follow the ethical principles of the Helsinki Declaration, the ethical regulations of China and the management norms and regulations of clinical research. The information related to this program and written informed consent must be submitted to the Ethics Committee, which can formally carry out the research only after obtaining written approval from the Ethics Committee. Researchers must submit annual reports to the Ethics Committee at least annually, if applicable. When the study is suspended and/or completed, the researcher must notify the Ethics Committee in writing; the researcher must report to the Ethics Committee in a timely manner the changes that have taken place in all the research work (such as the revision of the programme and/or informed consent).

#### 5. 2 informed consent

Informed consent may not be used until it has been approved

by the ethics committee. Before participating in this study, each subject or his legal representative should read the informed consent form and give him or her sufficient time to understand the details of this study after the detailed answers of the research doctor, so that the subjects or their legal representatives can be fully informed, and the subjects have the right to voluntarily choose whether to participate or follow up. The study was withdrawn at that time. Any modification of the informed consent must be approved by the ethics committee of the research hospital, and the patients without leaving the hospital must sign the new version of the informed consent. The informed consent shall be signed voluntarily by the subject himself or his legal representative. The informed consent signed by the researcher and the subjects themselves or their legal representatives is in duplicate and each party keeps one copy. Informed consent is kept for reference as an important document of clinical trials.

## 六、Cryptosecurity

- 1. The collection and processing of personal data of subjects selected for this study is limited to the data necessary for the purpose of this study. The information contained in the Research Institute (including data) is only provided to the project collaboration group for review. Without the approval of the project leader and the project collaboration group, it is strictly prohibited to provide any information to third parties unrelated to the study.
- 2. The project manager has the right to publish or publish information or data related to this test. If other individuals or units concerned with this test wish to publish or publish the test results or related data, they need to obtain the prior consent of the project leader. Project leaders should obtain the consent of researchers if they need to present the names of researchers in publications,

publications or advertisements.

## 七. Project participants

## 7.1 Research Institutes

 Research center: Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology

## -Collaboration unit:

| Number | Collaboration unit | Researcher |
|---|---|---|
| 1 | Anhui provincial hospital | Jia Weidong |
| 2 | China Meitan General Hospital | Li Tao |
| 3 | Beijing Tsinghua Changgeng<br>Hospital | Zeng Jianping |
| 4 | Beijing Tiantan Hospital<br>Affiliated to Capital Medical<br>University | Cheng Shi |
| 5 | Xuanwu Hospital, Capital Medical<br>University | Zheng Yamin |
| 6 | Beijing Youan Hospital Affiliated<br>to Capital Medical University | Zeng Daobing |
| 7 | General Hospital of the Chinese<br>People's Liberation Army | Wang Jing |
| 8 | Peking Union Medical College<br>Hospital | He Xiao Dong |
| 9 | Beijing Century Temple Hospital<br>Affiliated to Capital Medical<br>University | Peng Jirun |
| 10 | Zhongshan Hospital Affiliated to<br>Xiamen University | Su Yongjie |
| 11 | Zhangzhou Zheng Xing hospital | Li Jianguo |
| 12 | Union Medical College Hospital<br>Affiliated to Fujian Medical<br>University | Chen Yanling |
| 13 | First Affiliated Hospital of<br>Fujian Medical University | Zhang Zhibo |
| 14 | Meng Chao Liver and Gallbladder<br>Hospital of Fujian Medical<br>University | Zeng Yongyi |
| 15 | Second Hospital of Lanzhou<br>University | Cheng Zhibin |

| 16 | Foshan Chancheng District Central | |
|---|---|---|
| | Hospital | Peng Liang |
| 17 | Guangzhou First People's Hospital | Gu Weili |
| 18 | First Affiliated Hospital of<br>Shantou University | Yan Jiang |
| 19 | First Affiliated Hospital of<br>Shenzhen University | Zhan Yongqiang |
| 20 | Peking university shenzhen hospital | Liu Jikui |
| 21 | Sun Yat-sen University Cancer<br>Center | Li Shengping |
| 22 | Sun Yixian Memorial Hospital of<br>Sun Yat-sen University | Chen Yajin |
| 23 | Zhongshan People's Hospital | Chang Xiaojian |
| 24 | Affiliated Hospital of Guangdong Medical College | Chen Nianping |
| 25 | Guigang People's Hospital | Luo Hanchuan |
| 26 | Guiping People's Hospital | Wei Xiaoyuan |
| 27 | Liuzhou People's Hospital | Liu Qiang |
| 28 | First Affiliated Hospital of Guangxi Medical University | Peng Tao |
| 29 | Cancer Hospital Affiliated to Guangxi Medical University | Wu Feixiang |
| 30 | Guangxi Zhuang Autonomous Region<br>People's Hospital | Liu Tianqi |
| 31 | Sow District Hospital of traditional Chinese Medicine | Zhou Qiang |
| 32 | Danzhai County People's Hospital | Wang Huigang |
| 33 | Jinsha People's Hospital | Wang Changkuan |
| 34 | Liupanshui People's Hospital | Cheng Yongpeng |
| 35 | Tongren First People's Hospital | Zhu Yingqian |
| 36 | Xingyi People's Hospital | Peng Yanchun |
| 37 | People's Hospital of Xingyi City,<br>Guizhou Province | Luo Yunbo |
| 38 | Affiliated Hospital of Zunyi<br>Medical College, Guizhou Province | Liu Yao |
| 39 | Second Affiliated Hospital of<br>Guizhou Medical University (Kaili | |
| 40 | 418 Hospital) Affiliated Hospital of Guizhou Medical University | Shu Xiao<br>Sun Chengyi |

| 41 | Hainan Provincial People's | ZHENC I. C |
|---|---|---|
| | Hospital | ZHENG Jinfang |
| 42 | Affiliated Hospital of Hainan | Yang Yan |
| | Medical College | rang ran |
| 43 | Cangzhou Central Hospital | Li Xuefeng |
| 44 | The Fourth Hospital of Hebei | |
| | · | Peng Li |
| 45 | Hebi City People's Hospital, Henan | |
| | | Chang Yunfeng |
| 46 | People's Liberation Army 150 | |
| | Central Hospital | Sun Gaobin |
| 47 | Jingshan County People's Hospital, | Yang Yong |
| 10 | Hubei Province | |
| 48 | Fuyang City People's Hospital, | C D 1 |
| 40 | Henan Province | Gao Deshan |
| 49 | Tangyin County People's Hospital, | Car Clai |
| - FO | Henan Province | Su Shi |
| 50 | The First Affiliated Hospital of | Tang Zhe |
| F1 | Zhengzhou University | 71 |
| 51 | Henan Cancer Hospital | Zhou Jinxue |
| 52 | • | Han Yanhua |
| 53 | The Second Affiliated Hospital of | C. : V. |
| | - | Cui Yunyu |
| 54 | The Third Affiliated Hospital of Harbin Medical University (Tumor | |
| | Hospital) | Zhang Yubao |
| 55 | The Fourth Affiliated Hospital of | Zhang Tubao |
| 00 | Harbin Medical University | Xu Lishan |
| 56 | The First Affiliated Hospital of | Ad E13Hall |
| 30 | Harbin Medical University | Yin Dalong |
| 57 | Heilongjiang Provincial People's | |
| | Hospital | Jin Zhengxi |
| 58 | Jianghan Oilfield General Hospital | Zhang Yusheng |
| 59 | | Deng Youfa |
| 60 | Chongyang County People's Hospital | _ |
| 61 | | Deng Haibo |
| 62 | | Liu Baokuo |
| 63 | Daye City Hospital | Xiong Chunbo |
| 64 | Daye Nonferrous Pharmaceuticals | ATONG CHUNDO |
| 04 | Affiliated Hospital | Xu Ping |
| 65 | Dangyang People's Hospital | Xu Yuandeng |
| 55 | pandjand rechte a moshitar | na radiidelig |

| 66 | Ezhou Central Hospital | Chen Yifa |
|---|---|---|
| 67 | Enshi State Central Hospital | Li Jinmei |
| 68 | Gezhouba Central Hospital | Luo Jing |
| 69 | Public Security County People's<br>Hospital | Chen Houbin |
| 70 | Public Security County Hospital | Zou Xianxiong |
| 71 | Hanchuan People's Hospital | Yong Yongjun |
| 72 | Hong'an County People's Hospital | Gan Shenghong |
| 73 | Honghu People's Hospital | Li Ping |
| 74 | Honghu City Schistosomiasis<br>Specialist Hospital | Cao Yu |
| 75 | Union Hospital of Tongji Medical<br>College, Huazhong University of | Feng Xiansong |
| 76 | Huangpi District People's Hospital | Hu Yanjun |
| 77 | Huanggang Central Hospital | He Qianjin |
| 78 | Huanggang Chinese Medicine General<br>Surgery | Wang Xiao |
| 79 | Huangmei County People's Hospital | Wang Dahai |
| 80 | Huangmei County Chinese Medicine<br>Hospital | Yang Yuning |
| 81 | Huangshi Pu'ai Hospital | Shi Huxi |
| 82 | First Hospital of Huangshi City | Liu Xisong |
| 83 | Yellowstone Central Hospital | Xia Guobing |
| 84 | Huangzhou District People's<br>Hospital | Wang Jianguo |
| 85 | Jiayu County People's Hospital | Chen Yong |
| 86 | Jianli County People's Hospital | Yan Denggao |
| 87 | Jianshi County People's Hospital | Tang Liangqing |
| 88 | Jiangling County People's Hospital | Wang Qingshan |
| 89 | The 161st Hospital of the Chinese<br>People's Liberation Army | Xu Ke |
| 90 | | Li Wei |
| 91 | Jingzhou Central Hospital | Yang Zhiqi |
| 92 | Lichuan People's Hospital | Xiang Xianhui |
| 93 | Luotian County People's Hospital | Yu Shengfeng |
| 94 | Macheng Central Hospital | Yu Yiming |
| 95 | | Huang Ying |
| 96 | Hunchun County People's Hospital | Wang Zhirong |
| 97 | Qianjiang Central Hospital | Yin Tongzhi |

| Hospital 99 Luxi County People's Hospital Liu Fengshun 100 Songzi City People's Hospital He Qianzhang 101 Sui County People's Hospital Shen Tao 102 Suizhou Central Hospital Peng Gang 103 Tongshan County People's Hospital Cheng Shouren 104 Tuanfeng County People's Hospital Xu Shiying 105 Wuchang Railway Hospital Gao Xuzhong 106 Wuhan University People's Hospital Ding Youming 107 Zhongnan Hospital of Wuhan University 108 Wuhan Dongxihu Hospital You Jian 110 Hubei Rongjun Hospital Yang Guochao 111 Wuhan Sixth Hospital Liu Wen 112 Wuhan Xinzhou District People's Hospital 113 Wuhan Central Hospital Cai Changchun 114 Wuxue People's Hospital Cai Changchun 115 Lishui County People's Hospital Chen Xiaoming 116 Xiantao City People's Hospital Zeng Changjiang 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Hu Gioxing 110 Fuyang City Hospital of 121 Traditional Chinese Medicine Hu Bichuan 122 Xiaochang County People's Hospital Deng Xiaobin 123 Hubei Xinhua Hospital Hu Yongjun 124 Yangxin County People's Hospital Hu Yongjun 125 Yangxin County People's Hospital Hu Yongjun 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital 128 Yichang Central Hospital Huo Lei 127 Yiling District People's Hospital 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Cheng Jun 129 Yicheng People's Hospital Cheng Jun | 98 | National Pharmacy Dongfeng General | |
|---|---|---|---|
| 100 Songzi City People's Hospital He Qianzhang 101 Sui County People's Hospital Shen Tao 102 Suizhou Central Hospital Peng Gang 103 Tongshan County People's Hospital Cheng Shouren 104 Tuanfeng County People's Hospital Xu Shiying 105 Wuchang Railway Hospital Gao Xuzhong 106 Wuhan University People's Hospital Ding Youming 107 Zhongnan Hospital of Wuhan University He Yueming 108 Wuhan Dongxihu Hospital Cai Lie 109 Wuhan Puai Hospital You Jian 110 Hubei Rongjun Hospital Yang Guochao 111 Wuhan Sixth Hospital Liu Wen 112 Wuhan Xinzhou District People's Hospital Cai Changchun 114 Wuxue People's Hospital Ju Yiqing 115 Lishui County People's Hospital Chen Xiaoming 116 Xiantao City People's Hospital Zeng Changjiang 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County People's Hospital Hu Cuei 127 Yiling District People's Hospital 128 Yichang Second People Hospital Hu Lei 127 Yiling District People's Hospital 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Cheng Jun 129 Yicheng People's Hospital Cheng Jun | | | Zhou Wenbo |
| 101 Sui County People's Hospital Peng Gang 102 Suizhou Central Hospital Peng Gang 103 Tongshan County People's Hospital Cheng Shouren 104 Tuanfeng County People's Hospital Xu Shiying 105 Wuchang Railway Hospital Gao Xuzhong 106 Wuhan University People's Hospital Ding Youming 107 Zhongnan Hospital of Wuhan University Hey Yueming 108 Wuhan Dongxihu Hospital Cai Lie 109 Wuhan Puai Hospital You Jian 110 Hubei Rongjun Hospital Yang Guochao 111 Wuhan Sixth Hospital Liu Wen 112 Wuhan Xinzhou District People's Hospital 113 Wuhan Central Hospital Gai Changchun 114 Wuxue People's Hospital Ju Yiqing 115 Lishui County People's Hospital Chen Xiaoming 116 Xiantao City People's Hospital Zeng Changjiang 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Hu Yongjun 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Huo Lei 127 Yiling District People's Hospital 128 Yichang Second People Hospital 129 Yicheng People's Hospital Zheng Jun 129 Yicheng People's Hospital Cheng Jun 129 Yicheng People's Hospital | 99 | Luxi County People's Hospital | Liu Fengshun |
| 102 Suizhou Central Hospital Peng Gang 103 Tongshan County People's Hospital Cheng Shouren 104 Tuanfeng County People's Hospital Xu Shiying 105 Wuchang Railway Hospital Gao Xuzhong 106 Wuhan University People's Hospital Ding Youming 107 Zhongnan Hospital of Wuhan University 108 Wuhan Dongxihu Hospital Cai Lie 109 Wuhan Puai Hospital You Jian 110 Hubei Rongjun Hospital Liu Wen 111 Wuhan Sixth Hospital Liu Wen 112 Wuhan Xinzhou District People's Hospital Lu Jinxi 113 Wuhan Central Hospital Cai Changchun 114 Wuxue People's Hospital Ju Yiqing 115 Lishui County People's Hospital Zeng Changjiang 116 Xiantao City People's Hospital Hu Guoxing 118 Xianning First People's Hospital Liao Xiaofeng 119 Xiangyang Central Hospital Wang Daihong 110 Fuyang City Hospital Of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County People's Hospital Hu Cuei 127 Yiling District People's Hospital 128 Yichang Second People Hospital 129 Yicheng People's Hospital Zheng Jun 129 Yicheng People's Hospital Zheng Jun 129 Yicheng People's Hospital Cheng Jun 129 Yicheng People's Hospital Cheng Jun | 100 | Songzi City People's Hospital | He Qianzhang |
| Tongshan County People's Hospital Cheng Shouren 104 Tuanfeng County People's Hospital Xu Shiying 105 Wuchang Railway Hospital Gao Xuzhong 106 Wuhan University People's Hospital Ding Youming 107 Zhongnan Hospital of Wuhan University 108 Wuhan Dongxihu Hospital Cai Lie 109 Wuhan Puai Hospital Yang Guochao 110 Hubei Rongjun Hospital Liu Wen 111 Wuhan Sixth Hospital Liu Wen 112 Wuhan Xinzhou District People's Hospital Cai Changchun 113 Wuhan Central Hospital Gui Chen Xiaoming 116 Xiantao City People's Hospital Zeng Changjiang 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County People's Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 101 | Sui County People's Hospital | Shen Tao |
| 104 Tuanfeng County People's Hospital Xu Shiying 105 Wuchang Railway Hospital Gao Xuzhong 106 Wuhan University People's Hospital Ding Youming 107 Zhongnan Hospital of Wuhan University 108 Wuhan Dongxihu Hospital Cai Lie 109 Wuhan Puai Hospital You Jian 110 Hubei Rongjun Hospital Liu Wen 111 Wuhan Sixth Hospital Liu Wen 112 Wuhan Xinzhou District People's Hospital Cai Changchun 114 Wuxue People's Hospital Ju Yiqing 115 Lishui County People's Hospital Chen Xiaoming 116 Xiantao City People's Hospital Hu Guoxing 117 Xianning First People's Hospital Wang Daihong 118 Xianning Central Hospital Liao Xiaofeng 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County People's Hospital Huo Lei 127 Yiling District People's Hospital, 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 102 | Suizhou Central Hospital | Peng Gang |
| 105 Wuchang Railway Hospital 106 Wuhan University People's Hospital Ding Youming 107 Zhongnan Hospital of Wuhan University 108 Wuhan Dongxihu Hospital 109 Wuhan Puai Hospital 110 Hubei Rongjun Hospital 111 Wuhan Sixth Hospital 112 Wuhan Xinzhou District People's Hospital 113 Wuhan Central Hospital 114 Wuxue People's Hospital 115 Lishui County People's Hospital 116 Xiantao City People's Hospital 117 Xianning First People's Hospital 118 Xianning Central Hospital 119 Xiangyang Central Hospital 110 Fuyang City Hospital of 111 Traditional Chinese Medicine 112 Xiaochang County People's Hospital 113 Hubei Xinhua Hospital 114 Wang Daihong 115 Lishui County People's Hospital 116 Xianning First People's Hospital 117 Xianning First People's Hospital 118 Xianning Central Hospital 119 Xiangyang Central Hospital 110 Fuyang City Hospital of 111 Traditional Chinese Medicine 112 Xiaochang County People's Hospital 113 Hubei Xinhua Hospital 114 Yangxin County People's Hospital 115 Xiaogan Central Hospital 116 Xiaochang Second People Hospital 117 Xiaochang Second People Hospital 118 Xiaochang Central Hospital 119 Yichang Second People Hospital 110 Hue Viling District People's Hospital 111 Kubang Jun 112 Yichang Central Hospital 112 Yichang Central Hospital 113 Wang Vichang Central Hospital 114 Yichang Central Hospital 115 Liao Xiaochang Jun 116 Xiaochang Central Hospital 117 Xiaochang Jun 118 Xiaochang Central Hospital 119 Xiaochang Central Hospital 110 Hue Viling Jun 110 Hue Viling Jun 1110 Hue Viling Jun 110 Hue | 103 | Tongshan County People's Hospital | Cheng Shouren |
| 106 Wuhan University People's Hospital Ding Youming 107 Zhongnan Hospital of Wuhan University 108 Wuhan Dongxihu Hospital 109 Wuhan Puai Hospital 110 Hubei Rongjun Hospital 111 Wuhan Sixth Hospital 112 Wuhan Xinzhou District People's Hospital 113 Wuhan Central Hospital 114 Wuxue People's Hospital 115 Lishui County People's Hospital 116 Xiantao City People's Hospital 117 Xianning First People's Hospital 118 Xianning Central Hospital 119 Xiangyang Central Hospital 110 Fuyang City Hospital Of Traditional Chinese Medicine 120 Fuyang City Hospital Of Traditional Chinese Medicine 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital 123 Hubei Xinhua Hospital 124 Yangxin County People's Hospital 125 Yangxin County People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital 129 Yicheng People's Hospital 120 Ge Liang 121 Zheng Jun 122 Yichang Central Hospital 123 Zheng Jun 124 Yangxin County Hospital 125 Zheng Jun 126 Yichang Central Hospital 127 Yiling District People's Hospital 128 Yichang Central Hospital 129 Yicheng People's Hospital | 104 | Tuanfeng County People's Hospital | Xu Shiying |
| The Sunday and Hospital of Wuhan University 108 Wuhan Dongxihu Hospital 109 Wuhan Puai Hospital 110 Hubei Rongjun Hospital 111 Wuhan Sixth Hospital 112 Wuhan Xinzhou District People's Hospital 113 Wuhan Central Hospital 114 Wuxue People's Hospital 115 Lishui County People's Hospital 116 Xiantao City People's Hospital 117 Xianning First People's Hospital 118 Xianning Central Hospital 119 Xiangyang Central Hospital 120 Fuyang City Hospital of Traditional Chinese Medicine 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital 123 Hubei Xinhua Hospital 124 Yangxin County People's Hospital 125 Yangxin County People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital, Vichang City 128 Yichang Central Hospital 129 Yicheng People's Hospital 120 Ziang Central Hospital 121 Xiaochang Second People Hospital 122 Xiaogan Central Hospital 123 Yichang Central Hospital 124 Yangxin County Third People's 125 Yangxin County Third People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital 128 Yichang Central Hospital 129 Yicheng People's Hospital | 105 | Wuchang Railway Hospital | Gao Xuzhong |
| University 108 Wuhan Dongxihu Hospital 109 Wuhan Puai Hospital 110 Hubei Rongjun Hospital 111 Wuhan Sixth Hospital 112 Wuhan Xinzhou District People's Hospital 113 Wuhan Central Hospital 114 Wuxue People's Hospital 115 Lishui County People's Hospital 116 Xiantao City People's Hospital 117 Xianning First People's Hospital 118 Xianning Central Hospital 119 Xiangyang Central Hospital 110 Fuyang City Hospital Uiao Xiaofeng 120 Fuyang City Hospital Of Traditional Chinese Medicine 121 Xiaochang County People's Hospital Hu Guoxing 122 Xiaogan Central Hospital 123 Hubei Xinhua Hospital 124 Yangxin County People's Hospital 125 Yangxin County People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital, Vichang City 128 Yichang Central Hospital 129 Yicheng People's Hospital 120 Ziang Central Hospital 121 Xiaochang Second People Hospital 122 Xiaogan Central Hospital 123 Hubei Xinhua Hospital 124 Yangxin County Third People's Hospital 125 Yangxin County Third People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital 128 Yichang Central Hospital 129 Yicheng People's Hospital | 106 | Wuhan University People's Hospital | Ding Youming |
| 109 Wuhan Puai Hospital You Jian 110 Hubei Rongjun Hospital Yang Guochao 111 Wuhan Sixth Hospital Liu Wen 112 Wuhan Xinzhou District People's Hospital Lu Jinxi 113 Wuhan Central Hospital Cai Changchun 114 Wuxue People's Hospital Ju Yiqing 115 Lishui County People's Hospital Chen Xiaoming 116 Xiantao City People's Hospital Zeng Changjiang 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Hu Yongjun 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Huo Lei 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 107 | | He Yueming |
| 110 Hubei Rongjun Hospital 111 Wuhan Sixth Hospital 112 Wuhan Xinzhou District People's Hospital 113 Wuhan Central Hospital 114 Wuxue People's Hospital 115 Lishui County People's Hospital 116 Xiantao City People's Hospital 117 Xianning First People's Hospital 118 Xianning Central Hospital 119 Xiangyang Central Hospital 110 Fuyang City Hospital of Traditional Chinese Medicine 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital 123 Hubei Xinhua Hospital 124 Yangxin County People's Hospital 125 Yangxin County People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital 128 Yichang Central Hospital 129 Yicheng People's Hospital 120 Chen Xiaochang 121 Kiaochang County People's Hospital 122 Kiaogan Central Hospital 123 Hubei Xinhua Hospital 124 Yangxin County People's Hospital 125 Yangxin County Third People's 126 Yichang Second People Hospital 127 Yiling District People's Hospital 128 Yichang Central Hospital 129 Yicheng People's Hospital 129 Yicheng People's Hospital 129 Yicheng People's Hospital 120 Ge Liang | 108 | Wuhan Dongxihu Hospital | Cai Lie |
| 111 Wuhan Sixth Hospital 112 Wuhan Xinzhou District People's Hospital 113 Wuhan Central Hospital 114 Wuxue People's Hospital 115 Lishui County People's Hospital 116 Xiantao City People's Hospital 117 Xianning First People's Hospital 118 Xianning Central Hospital 119 Xiangyang Central Hospital 110 Fuyang City Hospital Of Traditional Chinese Medicine 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital 123 Hubei Xinhua Hospital 124 Yangxin County People's Hospital 125 Yangxin County People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital 129 Yicheng People's Hospital 120 Ge Liang 121 Zheng Jun 122 Zheng Jun 123 Hubei Xinhua Hospital 124 Yangxin County Third People's Hospital 125 Yangxin County Third People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital 128 Yichang Central Hospital 129 Yicheng People's Hospital 129 Yicheng People's Hospital 129 Yicheng People's Hospital 120 Ge Liang | 109 | Wuhan Puai Hospital | You Jian |
| Hospital Wuhan Xinzhou District People's Hospital Lu Jinxi Lu Jinxi Ruspital Wuhan Central Hospital Cai Changchun Lishui County People's Hospital Lishui County People's Hospital Lishui County People's Hospital Chen Xiaoming Chen Xiaoming Chen Xiaoming Zeng Changjiang Ruspital Liao Xiaofeng Namp Daihong Ruspital Hu Guoxing Ruspital Hu Bichuan Ruspital Hu Bichuan Ruspital Hu Bichuan Ruspital Hu Yongjun Ruspital Hu | 110 | Hubei Rongjun Hospital | Yang Guochao |
| Hospital 113 Wuhan Central Hospital 114 Wuxue People's Hospital 115 Lishui County People's Hospital 116 Xiantao City People's Hospital 117 Xianning First People's Hospital 118 Xianning Central Hospital 119 Xiangyang Central Hospital 120 Fuyang City Hospital of 121 Traditional Chinese Medicine 122 Xiaochang County People's Hospital 123 Hubei Xinhua Hospital 124 Yangxin County People's Hospital 125 Yangxin County People's Hospital 126 Yichang Second People Hospital 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital 129 Yicheng People's Hospital Tuy Yicheng People's Hospital Tuy Jing | 111 | Wuhan Sixth Hospital | Liu Wen |
| 114 Wuxue People's Hospital Ju Yiqing 115 Lishui County People's Hospital Chen Xiaoming 116 Xiantao City People's Hospital Zeng Changjiang 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Huo Lei 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City Yicheng People's Hospital Zheng Jun 128 Yicheng People's Hospital Ge Liang | 112 | - | Lu Jinxi |
| 115 Lishui County People's Hospital Chen Xiaoming 116 Xiantao City People's Hospital Zeng Changjiang 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Huo Lei 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City Zheng Jun 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 113 | Wuhan Central Hospital | Cai Changchun |
| 116 Xiantao City People's Hospital Zeng Changjiang 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Song Jinwen 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City Zheng Jun 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 114 | Wuxue People's Hospital | Ju Yiqing |
| 117 Xianning First People's Hospital Hu Guoxing 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Huo Lei 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 115 | Lishui County People's Hospital | Chen Xiaoming |
| 118 Xianning Central Hospital Wang Daihong 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Huo Lei 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 116 | Xiantao City People's Hospital | Zeng Changjiang |
| 119 Xiangyang Central Hospital Liao Xiaofeng 120 Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Song Jinwen 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 117 | Xianning First People's Hospital | Hu Guoxing |
| Fuyang City Hospital of Traditional Chinese Medicine Hu Bichuan 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 118 | Xianning Central Hospital | Wang Daihong |
| Traditional Chinese Medicine 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Huo Lei 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 119 | Xiangyang Central Hospital | Liao Xiaofeng |
| 121 Xiaochang County People's Hospital Deng Xiaobin 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Song Jinwen 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City Li Jianwen 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 120 | Fuyang City Hospital of | |
| 122 Xiaogan Central Hospital Hu Yongjun 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Song Jinwen 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Vichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | | Traditional Chinese Medicine | Hu Bichuan |
| 123 Hubei Xinhua Hospital Zhu Yixiang 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Song Jinwen 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City Li Jianwen 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 121 | Xiaochang County People's Hospital | Deng Xiaobin |
| 124 Yangxin County People's Hospital Ma Xianshi 125 Yangxin County Third People's Hospital Song Jinwen 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City Li Jianwen 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 122 | Xiaogan Central Hospital | Hu Yongjun |
| 125 Yangxin County Third People's Hospital 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Yichang City 128 Yichang Central Hospital 129 Yicheng People's Hospital Ge Liang | 123 | Hubei Xinhua Hospital | Zhu Yixiang |
| Hospital 126 Yichang Second People Hospital Huo Lei 127 Yiling District People's Hospital, Li Jianwen Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 124 | Yangxin County People's Hospital | Ma Xianshi |
| 127 Yiling District People's Hospital, Li Jianwen Yichang City 128 Yichang Central Hospital Zheng Jun 129 Yicheng People's Hospital Ge Liang | 125 | | Song Jinwen |
| Yichang City 128 Yichang Central Hospital 129 Yicheng People's Hospital Ge Liang | 126 | Yichang Second People Hospital | Huo Lei |
| 129 Yicheng People's Hospital Ge Liang | 127 | | Li Jianwen |
| | 128 | Yichang Central Hospital | Zheng Jun |
| | 129 | Yicheng People's Hospital | Ge Liang |
| 130 Yidu People's Hospital | 130 | Yidu People's Hospital | Hu Wen |
| 131 Yidu Chinese Medicine Hospital Yin Qinghua | 131 | Yidu Chinese Medicine Hospital | Yin Qinghua |

| 132 | Yingshan County People's Hospital | Shifeng |
|---|---|---|
| 133 | Yingcheng County People's Hospital | |
| 134 | Changyang County People's Hospital | Zhou Jigang |
| 135 | Changyang County Hospital of<br>Traditional Chinese Medicine | Yan Wandong |
| 136 | People's Liberation Army Wuhan<br>General Hospital | Lu Yuping |
| 137 | Zhongxiang People's Hospital | Su Jinsong |
| 138 | Hubei Cancer Hospital | Wu Dongde |
| 139 | Zigui County People's Hospital | Li Xuechun |
| 140 | Hunan Provincial People's Hospital | Mao Xianhai |
| 141 | Xiangxi People's Hospital | Wang Wener |
| 142 | Zhangpu County Chinese Medicine<br>Hospital | Xiang Jianwen |
| 143 | Huarong County People's Hospital | Wang Xuexiang |
| 144 | Central South University Xiangya<br>Hospital | Tang Huihuan |
| 145 | Zhuzhou Central Hospital | Tang Caixi |
| 146 | Baishen First Hospital of Jilin<br>University | Wang Guangyi |
| 147 | Jilin University Sino-Japanese<br>Friendship Hospital | Li Wei |
| 148 | Changzhou Third People's Hospital | Xu Locke |
| 149 | Nantong Cancer Hospital | Shao Bingfeng |
| 150 | Jiujiang City Duchang County<br>People's Hospital | Wang Longgang |
| 151 | Second Affiliated Hospital of<br>Nanchang University | Zou Shubing |
| 152 | The First Affiliated Hospital of<br>Nanchang University | Li Yong |
| 153 | The First Affiliated Hospital of Dalian Medical University | Wang Zhongyu |
| 154 | The First Affiliated Hospital of<br>Jinzhou Medical University | Bai Guang |
| 155 | Shenyang Military Region General<br>Hospital | Han Lei |
| 156 | Shengjing Hospital affiliated to<br>China Medical University | Wu Shuodong |
| 157 | Liaoning Cancer Hospital | Hua Xiangdong |
| 158 | The First Affiliated Hospital of<br>Inner Mongolia Medical University | Wang Zhenxia |

| 159 | Baotou Cancer Hospital | Zhao Qijun |
|---|---|---|
| 160 | | Bai Hua Tian |
| 161 | Ningxia Medical University General<br>Hospital | Yu Songning |
| 162 | Ningxia Hui Autonomous Region<br>People's Hospital | Li Mingwei |
| 163 | Affiliated Hospital of Qinghai<br>University | Fan Haining |
| 164 | Qinghai Provincial People's<br>Hospital | Guo Yamin |
| 165 | Qilu Hospital of Shandong<br>University | Zhixu Pavilion |
| 166 | Binzhou People's Hospital | Xia Xiuliang |
| 167 | Shan County Dongda Hospital | Li Hongsheng |
| 168 | Jining First People's Hospital | Jonson |
| 169 | Laiwu City People's Hospital | Zhao Zhiqiang |
| 170 | Shandong Provincial Hospital | Lu Jun |
| 171 | Liaocheng People's Hospital | Zhang Jinliang |
| 172 | Linyi Cancer Hospital | Li Enshan |
| 173 | Qingdao University Affiliated<br>Hospital | Wu Liqun |
| 174 | Qingdao Municipal Hospital | Shi Guangjun |
| 175 | Rizhao City Hospital | Xu Guixing |
| 176 | Yankuang Group General Hospital | Jiang Sifeng |
| 177 | Shanxi Grand Hospital | Zhao Haoliang |
| 178 | People's Liberation Army 323<br>Hospital | Yan Qimin |
| 179 | First Affiliated Hospital of Xi'an<br>Jiaotong University | Qi Zhimin |
| 180 | Renji Hospital, Shanghai Jiaotong<br>University School of Medicine | Wang Jian |
| 181 | Ruijin Hospital, Shanghai Jiao<br>Tong University School of Medicine | Han Tianquan |
| 182 | Xinhua Hospital, Shanghai Jiao<br>Tong University School of Medicine | Tang Zhaohui |
| 183 | Shanghai Tenth People's Hospital | Yin Lu |
| 184 | Zhongshan Hospital affiliated to<br>Fudan University | Liu Houbao |
| 185 | West China Hospital of Sichuan<br>University | Li Fuyu |

| 186 | Chengdu Military Region General | Tang Lijun |
|---|---|---|
| 105 | Hospital of Sichuan Province | |
| 187 | Deyang People's Hospital, Sichuan | 7 · |
| 1.00 | Province | Zeng Hui |
| 188 | Suining Central Hospital, Sichuan | D : V: |
| 100 | | Dai Yi |
| 189 | Zizhong County People's Hospital, | 71 01 |
| 100 | Sichuan Province | Zhuo Shijie |
| 190 | J 1 | Devotion |
| 191 | Tianjin Fourth Central Hospital | Wang Fengqi |
| 192 | Tianjin Nankai Hospital | Li Zhonglian |
| 193 | Tianjin Medical University Cancer<br>Hospital | Li Qiang |
| 194 | The First Affiliated Hospital of | |
| | Shihezi University Medical College | Peng Xinyu |
| 195 | Xinjiang Uygur Autonomous Region | |
| | Chinese Medicine Hospital | Duan Shaobin |
| 196 | Affiliated Tumor Hospital of | |
| | Xinjiang Medical University | Ding Wei |
| 197 | Xinjiang Uygur Autonomous Region | |
| | People's Hospital | Meng Hao 孟塬 |
| 198 | First Affiliated Hospital of | W . V . 1 |
| | Kunming Medical University | Wang Kunhua |
| 199 | Second Affiliated Hospital of | I : W - : |
| | Kunming Medical University | Li Weiming |
| 200 | Second Affiliated Hospital of | |
| | Zhejiang University School of | Li Jiangtao |
| | Medicine | |
| 201 | Hangzhou Normal University | D 71 · · · |
| | Affiliated Hospital | Pan Zhijian |
| 202 | Lishui Central Hospital, Zhejiang | |
| | Province | Tu Chaoyong |
| 203 | Zhejiang Yongjia Chinese Medicine | |
| | Hospital | Xie Dongmei |
| 204 | Daping Hospital of the Third | |
| | Military Medical University | Chen Ping |
| 205 | Third Military Medical University | |
| | - | Ding Shengcai |
| 206 | Southwest Military Hospital, Third | |
| | Military Medical University | Chen Zhiyu |
| 207 | | Zeng Jiangchao |

| 208 | Hepatobiliary Surgery, Chongqing | |
|-----|------------------------------------|---------------|
| | Emergency Medical Center | Liu Yongguo |
| 209 | Second Military Medical University | |
| | Eastern Hepatobiliary Surgery | |
| | Hospital | Zhang Yongjie |

#### 7.2List of researchers in the center

| Name | job title | division of work |
|---------------|-----------|------------------------------------------------|
| Wang Jianming | professor | overall plan |
| Tian Li | Doctor | Information collection, personnel coordination |
| Lu Yun | master | Information collection, personnel coordination |

#### 八. Reference

- [1] Hundal R, Shaffer E A. Gallbladder cancer: epidemiology and outcome[J]. Clin Epidemiol, 2014, 6(1):99-109.
- [2] Zou Shengquan, Zhang Lin. National Epidemiological Investigation Report on Gallbladder Cancer [J]. Chinese Journal of Practical Surgery, 2000, 20(1):43-46.
- [3] Cariati A, Andorno E. Cholesterol Gallstones Larger Than 3 cm Appear to be Associated With Gallbladder Cancer: Identification of an High Risk Group of Patients That Could Benefit From Preventive Cholecystectomy. [J]. Annals of Surgery, 2016, 263(3):e56.
- [4] Department of Biliary Surgery, Chinese Medical Association Surgery Branch. Guideline for the diagnosis and treatment of gallbladder cancer (2015)[J]. Chinese Journal of Digestive Surgery, 2015, 14(11):881-890.

- [5] Nakamura H, Arai Y, Totoki Y, et al. Genomic spectra of biliary tract cancer[J]. Nature Genetics, 2015, 47(9):1003.
- [6] Kanthan R, Senger JL, Ahmed S, Kanthan SC. Gallbladder Cancer in the 21st Century. J Oncol 2015;2015:967472.
- [7] Rakic M, Patrlj L, Kopljar M, Klicek R, Kolovrat M, Loncar B, Busic Z. Gallbladder cancer. Hepatobiliary Surg Nutr 2014;3:221-226.
- [8] Lee D G, Lee S H, Kim J S, et al. Loss of NDRG2 promotes epithelial-mesenchymal transition of gallbladder carcinoma cells through MMP-19-mediated Slug expression. [J]. Journal of Hepatology, 2015, 63(6):1429-1439.